CLINICAL TRIAL: NCT04479020
Title: REcanalization of Distal Cerebral Vessels in Acute Stroke Using ApeRio®
Status: Completed | Type: Observational
Sponsor: Acandis GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: REVISAR Revision 4.0
Record Dates: First submitted 2020-07-02; First posted 2020-07-21 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Acute Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Mechanical Thrombectomy — Mechanical thrombectomy requiring the use an APERIO® or APERIO® Hybrid(17) Thrombectomy device due to an thrombotic occlusion in a distal vessel of the anterior and posterior circulation (postbifurcal MCA, ACA, PCA)

SUMMARY:
The purpose of the REVISAR PMCF is to collect data in clinical practice of the APERIO® and APERIO® Hybrid(17) Thrombectomy Device, which are intended to restore blood flow in the neurovasculature by removing thrombus in patients experiencing ischemic stroke. Recanalization status will be assessed at the end of the procedure using the modified TICI (Thrombolysis in cerebral infarction) score.

DETAILED DESCRIPTION:
Study Type: prospective, multicenter, single-arm, open-label, national

Participants: 11 participating centers in Germany

PI: Dr. Franziska Dorn, University Hospital Bonn, Germany

Estimated Enrolment: A minimum of 130 patients treated with the APERIO® or APERIO® Hybrid(17) Thrombectomy Device due to thrombotic occlusions in a distal vessel of the anterior and posterior circulation (postbifurcal MCA, ACA, PCA)

Follow up: 3 months

Estimated Final Assessment: End of 2022

This is a prospective, multicenter, single-arm, open-label, national Post-Market Clinical Follow-up Study to collect comprehensive information on technical and clinical success and safety of the use of APERIO® and APERIO® Hybrid(17) Thrombectomy Device in a distal vessel of the anterior and posterior circulation (postbifurcal MCA, ACA, PCA). Aperio® and Aperio® Hybrid(17) Thrombectomy Device will be used within its approved indication.

ELIGIBILITY:
Inclusion Criteria:

* Any patient treated with the APERIO® or APERIO® Hybrid(17) Thrombectomy Device due to occlusion in distal vessel of the anterior and posterior circulation (postbifurcal MCA, ACA, PCA) according to IFU
* Age ≥ 18 years

Exclusion Criteria:

* pre stroke mRS ≥ 3
* Any contraindication according to IFU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with an APERIO® or APERIO® Hybrid(17) Thrombectomy Device due to a thrombotic occlusion in distal vessel of the anterior and posterior circulation (postbifurcal MCA, ACA, PCA).
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Primary efficacy endpoint | Immediatley after interventional procedure
  Successful arterial recanalization of occluded target vessel measured by mTICI score of 2b or 3 following the use of the APERIO® and APERIO® Hybrid(17) Thrombectomy Device without any symptomatic intracranial hemorrhage and rescue therapy within 3 passes per Device mTICI describes the response of thrombolytic therapy in ischemic stroke. Higashida et al. 2003: Grade 0: no perfusion Grade 1: penetration with minimal perfusion Grade 2: partial perfusion Grade 2A: only partial filling (less than two-thirds) of the entire vascular territory is visualized Grade 2B: complete filling of all of the expected vascular territory is visualized but the filling is slower than normal Grade 3: complete perfusion
Primary safety endpoint | 48 hours
  • Symptomatic intracranial hemorrhage (sICH): ICH in periprocedural (<48 hours) CT associated with worsening of NIHSS by ≥ 4 points within 48 hours.
Primary safety endpoint | 90 days
  Rates of device and procedure related (serious) adverse events ((S)AEs)
Primary Safety endpoint | 90 days
  Mortality

SECONDARY OUTCOMES:
Good neurological outcome | 90 days
  mRS (modified Ranking Scale)= 0-2
  0 No Symptoms
  1. No significant disability, despite symptoms, able to perform all usual duties and activities
  2. Slight disability; unable to perform all previous activities but able to look after own affairs without assistance
  3. Moderate disability; requires some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability bedridden incontinent and requires constant nursing care and attention
  6. Patient died

CONTACTS AND LOCATIONS:
Locations (11):
- Germany (11):
  - Schlosspark Klinik Charlottenburg, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Köln, Cologne
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Klinikum Fulda gAG, Fulda
  - Universitätsmedizin Göttingen, Göttingen
  - Universitätsklinikum des Saarlandes, Homburg
  - Universitätsklinikum Magdeburg A. ö. R., Magdeburg
  - Johannes Wesling Klinikum Minden, Minden
  - Klinikum der Universität München, München
  - radprax Neurozentrum Solingen, Solingen